CLINICAL TRIAL: NCT07407907
Title: The Effect of the Education Provided Based on the Information-Motivation-Behavioral Skills Model in Women Experiencing Hot Flashes During Menopause
Brief Title: Effect of IMB Model-Based Education for Women With Menopausal Hot Flashes
Acronym: IMB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Yeliz ILDIR ALTUN, Lecturer, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16.01.2024-06
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Menopausal Hot Flashes
Keywords: Menopause; Hot Flashes; Vasomotor Symptoms; Health Education; IMB Model; Quality of Life
MeSH Terms: conditions — Hot Flashes; Health Education

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an intervention group receiving IMB model-based education or a control group receiving no intervention. Both groups will be followed at baseline, 1 month, and 3 months after baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMB Model-Based Education Group (Experimental): A structured education program based on the Information-Motivation-Behavioral Skills (IMB) model was provided to women experiencing hot flashes during the menopausal period. The education program included information on the physiology of hot flashes, symptom management, lifestyle modifications, coping strategies, and the development of behavioral skills to manage menopausal symptoms.
  Interventions: Behavioral: IMB Model-Based Education Program
- Control Group (No Education) (No Intervention): This group consisted of women experiencing hot flashes during the menopausal period who did not receive any education or intervention during the study period. Participants continued their usual daily routines.

INTERVENTIONS:
Behavioral: IMB Model-Based Education Program — A structured education program based on the Information-Motivation-Behavioral Skills (IMB) model was delivered to women experiencing hot flashes during menopause. The intervention aimed to enhance participants' knowledge, motivation, and behavioral skills related to the management of menopausal hot flashes. The educational content included information on the physiology of hot flashes, lifestyle modifications, symptom management strategies, coping techniques, and skills to support healthy behaviors. The program was delivered through planned educational sessions.
  Arms: IMB Model-Based Education Group

SUMMARY:
This study was conducted to examine the effect of an education program based on the Information-Motivation-Behavioral Skills (IMB) Model on the level of hot flashes, overall menopausal symptoms, and quality of life in women experiencing hot flashes during the menopausal period.

The study consisted of an intervention group and a control group. The intervention group received a structured education program based on the IMB Model, while no education, counseling, or care intervention was provided to the control group. Both groups were assessed at baseline, and at the 1st and 3rd months following the intervention.

It is expected that the findings obtained from this study will demonstrate the effectiveness of IMB Model-based education in the management of menopausal vasomotor symptoms and contribute to the development of evidence-based nursing practices for women during the menopausal period.

ELIGIBILITY:
Inclusion Criteria:Women aged between 44 and 60 years.

Women in the perimenopausal or postmenopausal period.

A score of ≥ 10 on the Menopause-Specific Hot Flash Scale.

No diagnosis of severe chronic disease and no regular medication use related to such conditions.

Not receiving Hormone Replacement Therapy (HRT).

No diagnosed mental disorder requiring medical treatment.

Able to read, write, speak, and understand Turkish, with no language barriers.

Willingness to participate in the study and provision of voluntary informed consent.

-

Exclusion Criteria:Not meeting the inclusion criteria.

Initiation of Hormone Replacement Therapy during the study period.

Refusal to participate in the study.

Occurrence of an unexpected acute illness during the study period.

Withdrawal from the study at any stage by personal choice.

Incomplete completion of study questionnaires or forms after enrollment.

-

Ages: 44 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Hot Flash-Related Daily Interference | Baseline (pre-intervention), 1 month, and 3 months
  Hot flash-related daily interference was assessed using the Hot Flash Related Daily Interference Scale, which evaluates the extent to which hot flashes interfere with daily activities and quality of life.

SECONDARY OUTCOMES:
Hot Flush Beliefs | Baseline (pre-intervention), 1 month, and 3 months
  Hot flush-related beliefs were assessed using the Hot Flush Beliefs Scale (HFBS), which evaluates women's cognitive beliefs and perceptions related to hot flashes.
Menopause-Specific Quality of Life | Baseline (pre-intervention), 1 month, and 3 months
  Menopause-specific quality of life was assessed using the Menopause-Specific Quality of Life Scale, which evaluates the impact of menopausal symptoms on women's physical, psychological, and social well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice YILDIZ, Prof.Dr., Principal Investigator — Marmara University, Faculty of Health Sciences, Department of Obstetrics and Gynecology Nursing, Basıbuyuk RTE Health and Education Campus, 34854-Maltepe- Istanbul, Türkiye
Locations (1):
- Cumhuriyet University Health Services Application and Research Hospital, Obstetrics and Gynecology Outpatient Clinic, Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No